CLINICAL TRIAL: NCT05433844
Title: A Randomized, Open-label, Multiple-dose, Crossover Phase I Clinical Trial to Compare the Safety, Pharmacokinetics and Pharmacodynamics of JW0301 to C2105 in Healthy Subjects
Brief Title: To Evaluate the PK, PD, Safety and Drug Tolerance in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: JW21103
Record Dates: First submitted 2022-06-15; First posted 2022-06-27 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Intervention Model Description: A randomized, open, single-dose, 2x2 crossover-design clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Test Drug for Period I Reference Drug for Period II
  Interventions: Drug: Reference Drug or Test Drug
- Group 2 (Other): Reference Drug for Period I Test Drug for Period II
  Interventions: Drug: Reference Drug or Test Drug

INTERVENTIONS:
Drug: Reference Drug or Test Drug — Test Drug: single administration of JW0301 Reference Drug: single administration of C2105
  Tablet, Oral, QD for 1 Days, Washout period is more than 14 days after administration
  Other Names: Reference Drug(C2105) or Test Drug(JW0301)

SUMMARY:
1. To evaluate the pharmacokinetic and pharmacodynamics characteristics after administration of Reference Drug or Test Drug in healthy volunteers under fasting conditions
2. To evaluate the safety and drug tolerance after administration of Reference Drug or Test Drug in healthy volunteers under fasting conditions

DETAILED DESCRIPTION:
1. It is analyzed for subjects who receive scheduled clinical trial drugs according to the clinical trial plan, have no significant violations in comparative analysis, and have completed all scheduled blood collection for pharmacokinetic evaluation.

   To analyze subjects who receive clinical trial medications scheduled according to the clinical trial plan, have no significant violations in comparative analysis, and have assessable intragastric pH information by completing a 24-h pH monitoring measurement.
2. All subjects who received more than one dose of clinical trial drugs are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Subjects does not meet the Inclusion Criteria

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
AUCτ, SS(Area under the plasma drug concentration-time curve within a dosing interval at steady state) | 0 ~ 24h
  Evaluation PK for Esomeprazole after multiple dose
Percent decrease from baseline in integrated gastric acidity for 24-hour interval after 7th dose | Baseline versus Multiple dose during 7 days
  Evaluation PD for ambulatory 24hr pH monitor

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, PI, Principal Investigator — Clinical Trial Center, Seoul National University Hospital
Locations (1):
- Clinical Trial Center, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No